CLINICAL TRIAL: NCT05584397
Title: Comparing Immune Activation and Latent HIV Reservoir Size Between People Living With HIV (PWH) on Tenofovir-containing Versus NRTI-sparing ART
Brief Title: Comparing Immune Activation and Latent HIV Reservoir Size Between People Living With HIV on Tenofovir-containing Versus NRTI-free ART
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, German Gornalusse, Acting Assistant Professor, School of Medicine, OBGYN, University of Washington
Other Study IDs: STUDY00011699; R01AI134293 (NIH); KL2TR002317 (NIH)
Record Dates: First submitted 2022-10-05; First posted 2022-10-18 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: HIV-1-infection; HIV Disease Progression; Inflammation; HIV
Keywords: HIV reservoir; Interferon Stimulated Genes; Tenofovir; Interferon; Duodenum; Blood; Rectum; NRTI
MeSH Terms: conditions — Inflammation | interventions — Phlebotomy; Proctoscopy; Endoscopy, Digestive System; Gastroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood obtained from venipuncture during the first (screening) visit will be used to test for: 1) HIV plasma viral load; 2) peripheral blood CD4+ T cell count; 3) complete blood count (CBC); 4) prothrombin time (PT) and partial thromboplastin time (PTT); 5) and renal (kidney) function. Blood obtained from venipuncture during the second (procedure) visit will be used for RNA studies and PBMC and plasma isolation and storage. Biopsy samples (a total of 5 per site) will be isolated from the rectum and duodenum, by anoscopy and esophagogastroduodenoscopy (EGD), respectively. In both cases (anoscopy and EGD), samples will be preserved in RNAlater (for RNA and DNA analysis and potentially immunohistology) and some biopsies may be dry frozen (for potential proteomics study and determination of drug levels). Cytobrush samples will also be collected from both rectum and duodenum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tenofovir-containing ART: Cohort 1: Tenofovir-containing ART (tenofovir disoproxil fumarate [TDF] OR tenofovir alafenamide [TAF] PLUS any other ART drugs) prescribed for daily use by participants' primary care providers.
  Interventions: Procedure: Venipuncture; Procedure: Targeted physical medical exam; Procedure: Urine pregnancy test; Procedure: Anoscopy; Procedure: Esophagogastroduodenoscopy (EGD)
- NRTI-sparing ART: Cohort 2: NRTI-sparing ART (specifically: rilpivirine PLUS dolutegravir OR rilpivirine PLUS cabotegravir) prescribed for daily use by participants' primary care providers.
  Interventions: Procedure: Venipuncture; Procedure: Targeted physical medical exam; Procedure: Urine pregnancy test; Procedure: Anoscopy; Procedure: Esophagogastroduodenoscopy (EGD)

INTERVENTIONS:
Procedure: Venipuncture — Draw of peripheral blood (about 20 ml and 40 ml, during the screening and procedure visits, respectively).
  Other Names: Peripheral blood draw by phlebotomy
Procedure: Targeted physical medical exam — Study participants will be undergoing a physical exam where vitals will be recorded (e.g. temperature, blood pressure, heart rate). The registered nurse (RN) will also perform auscultation of heart and lungs.
  Study participants will be also asked to fill out a survey with questions related to his/her medical history, current use of medications, sexual history and substance abuse.
Procedure: Urine pregnancy test — Women of childbearing potential will be asked to run an urine pregnancy test during the second (procedure) visit. Pregnant women will not be allowed to participate in the study.
Procedure: Anoscopy — The anoscopy is an examination using a small, rigid, tubular instrument called anoscope (also called an anal speculum). This is inserted a few inches into the rectum in order to collect some small samples of mucosal tissue. We will collect 5 rectum biopsy samples and one cytobrush.
Procedure: Esophagogastroduodenoscopy (EGD) — The EGD involves looking at the esophagus, stomach, and first and second portion of the duodenum. This procedure involves the use of an endoscope to remove small tissue samples. This procedure uses conscious sedation drugs given by a vein in the arm. The procedure takes about 1½-2 hours, including time for recovery. We will collect 5 duodenal biopsies and one cytobrush.
  Other Names: Upper endoscopy

SUMMARY:
The goal of the project is to determine the difference in immune activation and HIV reservoir size between People living with HIV (PWH) on tenofovir-containing antiretroviral therapy (ART) versus PWH on nucleoside reverse transcriptase inhibitor (NRTI)-sparing ART. Tenofovir (TFV), a phosphonated nucleoside reverse transcriptase inhibitor (NRTI), is being used for oral pre-exposure prophylaxis (PrEP).

The investigators will test this hypothesis: tenofovir, and perhaps NRTIs in general, stimulate a type I/III interferon also in PWH who take these drugs. Because chronic interferon stimulation may promote the survival and proliferation of cells with integrated provirus, the investigators also hypothesize that these drugs antagonize decay of the HIV latent reservoir in PWH on ART. Consequently, the researchers hypothesize that PWH who have switched from NRTI-containing ART to NRTI-sparing ART exhibit lower type I/III interferon pathway activation and lower latent HIV reservoir size.

The investigators also hypothesize that independently of treatment, the extent of type I/III interferon activation correlates with latent HIV reservoir size.

Thus, the proposed study seeks to answer these two questions. Can the gastrointestinal epithelium be impacted by ART, and contribute to chronic immune activation and expansion of the HIV-1 reservoir? If so, what therapeutic approaches can the investigators implement to reduce the HIV-1 proviral load? The data will reveal pathways that can be targeted therapeutically to treat chronic immune activation in PWH. The findings of this study will immediately translate to optimize the standard of care in PWH.

DETAILED DESCRIPTION:
The study will be open-label, cross-sectional, two-cohort study (20 participants per cohort will be recruited).

Cohort 1: Tenofovir-containing ART (tenofovir disoproxil fumarate [TDF] OR tenofovir alafenamide [TAF] PLUS any other ART drugs) prescribed for daily use by participants' primary care providers.

Cohort 2: NRTI-sparing ART (specifically: rilpivirine PLUS dolutegravir OR rilpivirine PLUS cabotegravir) prescribed for daily use by participants' primary care providers.

The investigators plan to test type I/III IFN (interferon) pathway activation using Crystal digital PCR (Crystal-dPCR) to quantify mRNA copy numbers of ISG15 (ISG15 ubiquitin-like modifier), MX1 (MX dynamin like GTPase 1) and IFI6 (interferon alpha inducible protein 6). RNA will be isolated from the rectal and duodenal biopsies stored in RNALater using the RNeasy Fibrous Tissue Mini Kit (Qiagen) and from the PBMC using the RNeasy Plus Mini Kit (Qiagen). Crystal-dPCR will be performed on a 6-color Naica Crystal digital PCR instrument (Stilla Technologies).

The latent HIV reservoir will be measured in DNA derived from peripheral blood mononuclear cells (PBMCs) using a novel intact/defective proviral HIV DNA Crystal-dPCR assay developed jointly by the Hladik and Jerome groups in Seattle.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV infection, by two different positive antibody tests and/or detectable plasma HIV RNA on two different dates
2. ≥18 and ≤65 years of age
3. Stable use of ART medication for ≥ 1 year
4. No switch of ART regimen within the past 180 days
5. CD4 > 350/mm3 within the past 180 days
6. HIV RNA <40 copies / mL on ≥ 2 occasions during continuous ART of ≥ 1 years, with no blip of >1000 HIV RNA copies / mL
7. Karnofsky score ≥80
8. Willingness and ability to provide informed consent for study participation
9. Willingness to undergo all required study procedures

Exclusion Criteria:

1. Active malignancy including myelodysplastic syndrome, or myeloproliferative disease within 24 weeks prior to study entry
2. Prior organ or bone marrow transplantation
3. Diagnosed autoimmune disease
4. Medical need for ongoing treatment with an immunosuppressive drug
5. Diagnosis of AIDS (defined as any AIDS-defining opportunistic infection or cancer, or a history of blood CD4+ T cell count < 200/μL)
6. Active opportunistic infection
7. Vomiting or diarrhea which prohibits consistent use of ART
8. Pregnant or breastfeeding
9. Excessive ingestion of ethanol determined by an AUDIT score of >8
10. Substance abuse
11. History of medical non-compliance
12. The following laboratory values (< 30 days before enrollment):

    * Hemoglobin < 8.5 mg/dL
    * Platelet count < 100,000/μL
    * Coagulation (PT/PTT) tests above the normal reference
    * Creatinine clearance < 60 mL/min
13. Using disallowed medications:

    * Systemic corticosteroids
    * Other immunosuppressive medications (e.g., cyclosporine, sirolimus, tacrolimus, pimecrolimus, tofacitinib)
14. BMI > 40
15. Pulmonary dysfunction.
16. Use of narcotics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with HIV (PWH) on stable use of antiretroviral therapy (ART). They will be between 18 and 65 years of age. Children less than 18 years of age are excluded. Women of childbearing potential should not be pregnant to participate.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Type I/III Interferon pathway activation | Biopsy samples to assess interferon pathway activation will be collected during surgery. The assessment of this outcome (the determination of mRNA copy number) will be done around within one year of completing sample collection.
  Quantification of the mRNA copy number of the following Interferon-Stimulated Genes (ISGs): ISG15 (ISG15 ubiquitin-like modifier), MX1 (MX dynamin-like GTPase 1) and IFI6 (interferon alpha inducible protein 6). Copy numbers will be determined by Crystal digital PCR (dPCR), using the levels of UBC (Ubiquitin C) mRNA copies as normalizers.
Size of the latent intact proviral HIV reservoir in cell-associated HIV DNA (Ca-DNA) | Blood samples to assess the latent HIV reservoir will be collected during surgery. The assessment of this outcome (the determination of HIV copy number) will be done around within one year of completing sample collection.
  Determination of size (copy number) of the HIV proviral intact reservoir using a recently published assay the Hladik's lab conjointly with Jerome's lab developed (reference: Levy et al., 2021, Cell Reports Medicine 2, 100243). This outcome will be expressed as intact HIV copy numbers (found in cell-associated HIV DNA) per 10^6 T cells. We will use a multiplexed digital PCR (dPCR) assay that simultaneously quantifies likely intact HIV-1 proviruses and T lymphocytes. We designed two triplex droplet digital PCR assays, each with 2 unique targets and 1 in common, and normalize the results to PCR-based T cell counts. Both HIV assays are specific, sensitive, and reproducible. Together, they estimate the number of proviruses containing all five primer-probe regions.
Size of the latent defective proviral HIV reservoir in cell-associated HIV DNA (Ca-DNA) | Blood samples to assess the latent HIV reservoir will be collected during surgery. The assessment of this outcome (the determination of HIV copy number) will be done around within one year of completing sample collection.
  Determination of size (copy number) of the HIV proviral defective reservoir using a recently published assay the Hladik's lab conjointly with Jerome's lab developed (reference: Levy et al., 2021, Cell Reports Medicine 2, 100243). This outcome will be expressed as defective HIV copy numbers (found in cell-associated HIV DNA) per 10^6 T cells.

SECONDARY OUTCOMES:
Composition of gastrointestinal microbiota | Cytobrush samples to assess gut microbiota will be collected during surgery. The assessment of this outcome (the determination of 16s repertoire) will be done around within one year of completing sample collection.
  We will do 16s RNA sequencing in rectum and duodenum cytobrush samples to identify, classify and quantify gut microbiota.

OTHER OUTCOMES:
Determination of proteins that are secreted in the rectum and duodenum | Cytobrush samples to assess secreted proteins will be collected during surgery. The assessment of this outcome (the determination of the proteome) will be done around within one year of completing sample collection.
  We will conduct an unbiased proteomics approach to characterize the proteins that are secreted in both duodenum and rectum.
Determination of the global transcriptome | Blood and biopsy samples will be collected during surgery. The assessment of this outcome (the characterization of the transcriptome will be done around within one year of completing sample collection.
  We will do global transcriptomics analysis using sequencing of biopsy and blood mRNA

CONTACTS AND LOCATIONS:
Overall Officials: German G Gornalusse, PhD, MSc, Principal Investigator — University of Washington; Florian Hladik, MD, PhD, Principal Investigator — University of Washington; Romel D Mackelprang, PhD, MSc, Principal Investigator — University of Washington
Locations (1):
- University of Washington Positive Research and the Gastroenterology Clinic at Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We may share information encompassing global transcriptome analysis (e.g. RNA-Seq data) derived from biopsy or peripheral blood mononuclear cells (PBMC) mRNA, DNA sequencing of the bacterial 16S RNA gene from cytobrush material (to determine microbial composition in duodenum or rectum) and HIV proviral sequencing (to characterize the HIV reservoir). HIV status and the size/structure of the HIV reservoir will be data that will be shared. Direct identifiers (e.g., names, telephone numbers, emails, social security numbers, medical record numbers, etc.) will not be shared. Data will be submitted to the National Institute of Health (NIH) Genomic Data repository, with unrestricted access (i.e. data will be made accessible to anyone via a public website). The data will be coded or anonymized prior to submission to NIH such that the identities of subjects cannot be readily ascertained or otherwise associated with the data by the repository staff or secondary data users.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be shared at the time of submission of the scientific paper(s).
Access Criteria: The information from this study will be stored in a public unrestricted data bank that anyone can use. The National Institutes of Health (NIH) has developed data banks that collect genomic study data. The NIH will store the de-identified information in these data banks for other researchers to use in future studies on any topic. This will include de-identified information about the participants' HIV status, mRNA sequences or genomic allelic variants (e.g. single nucleotide polymorphisms and copy number variants). The researchers could be from government, academic, or commercial institutions. We have a Extramural Institutional Certification dated 01/07/2022, Genomic Program Administrator: Chris Marcus from the National Institute of Allergy and Infectious Diseases (NIAID), NIH, HHS.

REFERENCES:
- [Background] Hughes SM, Levy CN, Calienes FL, Stekler JD, Pandey U, Vojtech L, Berard AR, Birse K, Noel-Romas L, Richardson B, Golden JB, Cartwright M, Collier AC, Stevens CE, Curlin ME, Holtz TH, Mugo N, Irungu E, Katabira E, Muwonge T, Lama JR, Baeten JM, Burgener A, Lingappa JR, McElrath MJ, Mackelprang R, McGowan I, Cranston RD, Cameron MJ, Hladik F. Treatment with Commonly Used Antiretroviral Drugs Induces a Type I/III Interferon Signature in the Gut in the Absence of HIV Infection. Cell Rep Med. 2020 Sep 22;1(6):100096. doi: 10.1016/j.xcrm.2020.100096. PMID 33015651

DOCUMENTS (2):
  • Study Protocol (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT05584397/Prot_000.pdf
  • Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT05584397/ICF_001.pdf